CLINICAL TRIAL: NCT00932555
Title: EffeKt Taiwan- Efficacy and Safety of Long-term Treatment With KOGENATE® FS in Taiwan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Taiwan LTD
Other Study IDs: 14344; KG0803 (Other: company internal)
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Hemophilia A
Keywords: Octocog alfa; Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222)

INTERVENTIONS:
Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Patients under daily life treatment receiving Kogenate according to local drug information.

SUMMARY:
The aim of this international prospective post-marketing surveillance study is to obtain data on treatment procedures, long-term safety and efficacy and patient acceptance of KOGENATE Bayer/FS in treatment of patients with haemophilia A under daily-life treatment conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of hemophilia A, independent of age, treated with KOGENATE FS as their only source of FVIII, decision taken by the investigator to administer KOGENATE FS. For pretreated patients with more than 100 exposure days an inhibitor assessment within three months prior to enrollment should be available; for pretreated patients with less than 100 exposure days an inhibitor assessment at baseline should be available.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients with a diagnosis of hemophilia A. Physicians should consult the full prescribing information for KOGENATE® FS before enrolling patients and familiarize themselves with the safety information in the product package label.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2009-04; Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Efficacy and Safety of Kogenate FS | After 12 months and after 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Taiwan